CLINICAL TRIAL: NCT00429351
Title: Aromatic Amino Acid Metabolism in the Pathogenesis of Kwashiorkor
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Farook Jahoor, Professor, Pediatrics-Nutrition, Baylor College of Medicine
Other Study IDs: H-16233; R01DK075018 (NIH)
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Kwashiorkor
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, expired breath

SUMMARY:
This research may explain whether a shortage of three special compounds called aromatic amino acids is responsible for the severe illness and high death rate of children with the kwashiorkor type of malnutrition and whether supplying adequate amounts of these compounds in the treatment diet will speed up recovery from this condition. We propose that decreased availability of the aromatic amino acids may be the reason why children with kwashiorkor are sicker and more difficult to treat.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished children between 6 to 18 months of age.
* To standardize for degree of malnutrition, only patients whose weight is < 80 % of that expected for age will be enrolled. By the Wellcome Classification (22), enrolled patients will have marasmus (< 60 % weight/age and no edema), marasmic-kwashiorkor (< 60 % weight/age plus edema) or kwashiorkor (< 80 % weight/age plus edema).
* Presence of infection at admission. Infection will be defined by the presence of two or more of the following: Leukocyte count >11,000 cells/dl, temperature at admission > 99 oF, positive blood or urine cultures.

Exclusion Criteria:

* Criteria for exclusion will include presence of cardiovascular, hepatic, renal, gastrointestinal, metabolic disease or HIV/AIDS.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 82 children aged 6 to 18 months and diagnosed with severe protein-energy malnutrition. By the Wellcome Classification patients will have marasmus (< 60 % weight/age and no edema), marasmic-kwashiorkor (< 60 % weight/age plus edema) or kwashiorkor (< 80 % weight/age plus edema)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2006-09; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical Metabolism Research Unit, University of the West Indies, Mona, Kingston, Jamaica